CLINICAL TRIAL: NCT04160767
Title: Celiac Disease and Vitamin Status: Evaluation of the Effect of Supplementation With a Probiotic (VIVOMIXX®) on Vitamin B6, B12, 25'OH D, Folic Acid and Omocystein Levels, Metabolic and Inflammatory Status, and Gut Microbiota Metabolomics in a Cohoort of Celiac Patients
Brief Title: Celiac Disease and Vitamin Status: Evaluation of the Effect of Supplementation With a Probiotic (VIVOMIXX®) in a Cohoort of Celiac Patients
Acronym: VIVOMIXX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Elvira Verduci, Principal Investigator, Paediatrician, University of Milan Researcher, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015/ST/135-3
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Gut microbiota
MeSH Terms: conditions — Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator)
  Interventions: Drug: Probiotic Vivomixx; Behavioral: Gluten free diet
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Gluten free diet; Other: Placebo

INTERVENTIONS:
Drug: Probiotic Vivomixx — VIVOMIXX once a day for 4 months. VIVOMIXX® is a probiotic containing 8 differenct strains of bacteria: Streptococcus thermophilus DSM 24731, bifidobacteria (B. breve DSM 24732, B. longum DSM 24736, B. infantis DSM 24737) lactobacilli (L. acidophilus DSM 24735, L. plantarum DSM 24730, L. paracasei DSM 24733, L. delbrueckii subsp. bulgaricus DSM 24734). Every sachet contains 450 billions of bacteria, maltose and silicon dioxide. VIVOMIXX® will be freely given by the society MENDES S.A. - Lugano Switzerland.
  Arms: Probiotic
Behavioral: Gluten free diet — Gluten free diet will be encouraged in both arms
Other: Placebo — Placebo with same taste than VIVOMIXX, containing maltose and silicon dioxide once a day for 4 months.
  Arms: Placebo

SUMMARY:
Celiac disease is a disorder caused by a disregulation of the immune system which leads to immune response to gluten. Diet therapy is the gold standard of treatment, and the only effective one. Macronutrients and micronutrients deficiency (vitamin D, folic acid, vitamin B12, vitamin B6, iron and zinc), which is in any case far more common in patients who don't follow gluten free diet, can persist in a subset of patients who follow gluten-free diet. Supplementation of vitamins in these patients may have a beneficial role. A recent study in a murine model showed that supplementation with probiotic VIVOMIXX® leads to an increase in expression of vitamin D receptors in proximal and distal colon.

This is an interventional controlled randomized double blind study, which evaluates the effect of VIVOMIXX® on vitamin status.

DETAILED DESCRIPTION:
90 patients with celiac disease who follow gluten free diet will be enrolled. INCLUSION CRITERIA

* Celiac disease (diagnosis made according to ESPGHAN criteria) EXCLUSION CRITERIA
* Supplementation with pre/probiotics in the previous 3 months;
* Antibiotic therapy in the previous 3 months;
* Comorbidity with other acute (in the previous 3 months) or chronic gastrointestinal disorders
* Supplementation with group B vitamins for any reason

Patients enrolled will be referred to Paediatric Gastroenterology Service in San Paolo Hospital at the time of enrollement (T0) and after intervention therapy (T1, + 4 months).

Patients will be randomized in one of the two arms of intervention (VIVOMIXX once a day for 4 months versus placebo once a day for 4 months).

VIVOMIXX® is a probiotic containing 8 differenct strains of bacteria: Streptococcus thermophilus DSM 24731, bifidobacteria (B. breve DSM 24732, B. longum DSM 24736, B. infantis DSM 24737) lactobacilli (L. acidophilus DSM 24735, L. plantarum DSM 24730, L. paracasei DSM 24733, L. delbrueckii subsp. bulgaricus DSM 24734). Every sachet contains 450 billions of bacteria, maltose and silicon dioxide. VIVOMIXX® will be freely given by the society MENDES S.A. - Lugano Switzerland.

At each time point clinic evaluation, nutritional assessment and blood testing will be made. Data collection will include:

* Systemic arterial blood pressure;
* Anthropometric measures (height, weight, body mass index, waist circumference, triceps skinfold)
* Clinical evaluation including presence/absence of oral aphtous stomatitis
* Measure of chinolinic acid, serotonin, ghrelin (analysis will be made at Istituto Malattie Infettive, Università La Sapienza, Roma).
* Dosing of inflammatory markers (analysis will be made at Health Sciences Department, San Paolo Hospital).
* Metabolomics on stool samples (analysis will be made at Bologna University, Dipartimento di Scienze e Tecnologie Agro-Alimentari, Cesena, with a financial fund by MENDES S.A. - Lugano Switzerland).
* Routine blood testing including complete blood cell count, vitamin B6, acid folic, vitamin B12, vitamin D 25'OH, fasting glucose, fasting insulin, total cholesterol, LDL and HDL cholesterol, Apolipoprotein A1 and Apolipoprotein B, triglycerides, homocistein, auto-antibody anti endomisium and anti-transglutaminase,
* Genetic testing for MTHFR gene
* ESR, highly sensitive CRP, IL6, TNFalfa, fibrinogen
* Fecal calprotectin.

ELIGIBILITY:
Inclusion Criteria:

* Celiac disease (diagnosis made according to European Society for Paediatric Gastroenterology Hepatology and Nutrition)

Exclusion Criteria:

* Supplementation with pre/probiotics in the previous 3 months;
* Antibiotic therapy in the previous 3 months;
* Comorbidity with other acute (in the previous 3 months) or chronic gastrointestinal disorders
* Supplementation with group B vitamins for any reason

Max Age: 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Changes in vitamin B6, folic acid, vitamin B12 and 25'OH vitamin D levels in blood | Time point 0: day 0 Time point 1: after 4 months
Changes in homocysteine levels in blood | Time point 0: day 0 Time point 1: after 4 months
Changes in ghrelin, chinolinic acid and serotonin levels | Time point 0: day 0 Time point 1: after 4 months
Changes in fecal metabolomics (including production of short chain fatty acids verified by gas-chromatography) | Time point 0: day 0 Time point 1: after 4 months
Changes in highly sensitive C reactive protein levels | Time point 0: day 0 Time point 1: after 4 months
Changes in erythrocite sedimentation rate | Time point 0: day 0 Time point 1: after 4 months
Changes in fibrinogen blood levels | Time point 0: day 0 Time point 1: after 4 months
Changes in IL-6 blood levels | Time point 0: day 0 Time point 1: after 4 months
Changes in Tumor Necrosis Factor alfa blood levels | Time point 0: day 0 Time point 1: after 4 months

SECONDARY OUTCOMES:
Changes in body mass index | Time point 0: day 0 Time point 1: after 4 months
Changes in systemic arterial systolic and diastolic blood pressure | Time point 0: day 0 Time point 1: after 4 months
Changes in height | Time point 0: day 0 Time point 1: after 4 months
Changes in weight | Time point 0: day 0 Time point 1: after 4 months
Changes in waist circumference | Time point 0: day 0 Time point 1: after 4 months
Entity of reduction of triceps skinfold thickness | Time point 0: day 0 Time point 1: after 4 months
Changes in prevalence of aphtous stomatitis | Time point 0: day 0 Time point 1: after 4 months
Changes in chinolinic acid, serotonin, ghrelin levels in blood | Time point 0: day 0 Time point 1: after 4 months
Changes in complete cell blood count | Time point 0: day 0 Time point 1: after 4 months
Changes in total cholesterol levels | Time point 0: day 0 Time point 1: after 4 months
Changes in HDL cholesterol levels | Time point 0: day 0 Time point 1: after 4 months
Changes in LDL cholesterol levels | Time point 0: day 0 Time point 1: after 4 months
Changes in triglycerides levels | Time point 0: day 0 Time point 1: after 4 months
Changes in Apolipoprotein A1 levels | Time point 0: day 0 Time point 1: after 4 months
Changes in Apolipoprotein B levels | Time point 0: day 0 Time point 1: after 4 months
Changes in fasting glucose levels | T0 T1 (+4 months)
Changes in fasting insulin levels | Time point 0: day 0 Time point 1: after 4 months
Changes in auto-antibody anti endomisium titer | Time point 0: day 0 Time point 1: after 4 months
Changes in auto-antibody anti-transglutaminase titer | Time point 0: day 0 Time point 1: after 4 months
Changes in fecal calprotectin levels | Time point 0: day 0 Time point 1: after 4 months
Prevalence of wildtype allele of MTHFR gene by gene sequencing | Time point 0: day 0 (at the enrollement)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Paolo, Milan, Italy

IPD SHARING:
Plan to Share IPD: No